CLINICAL TRIAL: NCT03842722
Title: Insufficient Oxygenation in Septic Patients
Acronym: INOX-SEPSIS
Status: Completed | Type: Observational
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.G. van der Bom, Manager clinical transfusion research, Leiden University Medical Center
Other Study IDs: NL64824.058.18
Record Dates: First submitted 2018-10-22; First posted 2019-02-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Critical Care; Mitochondria; Oxygen; Fluid Therapy
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken for measurement of: creatinine, hemoglobin, lactate, central venous oxygen saturation, arterial saturation, arterial oxygen tension, venous oxygen tension, central venous-to-arterial carbon dioxide partial pressure difference. Furthermore, blood based cellular function will be assessed (presence of reactive oxygen species molecules, mitochondrial membrane potential and glutathione activity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill septic patients: Cohort: patients admitted via the emergency department or hospital ward to the intensive care unit of Leiden University Medical Center with the diagnosis sepsis or septic shock, who receive fluid therapy (either colloid, crystalloid and/or red blood cell) in their first day of admission to the ICU.
  Interventions: Device: Protoporphyrin IX - Triplet State Lifetime Technique

INTERVENTIONS:
Device: Protoporphyrin IX - Triplet State Lifetime Technique — Protoporphyrin IX - Triplet State Lifetime Technique is a way to measure mitochondrial oxygen tension in a non-invasive way at bedside.

SUMMARY:
This study will describe the change of mitochondrial oxygen tension (mitoPO2) compared to traditional parameters of oxygenation and oxygen balance in the first 24 hours of septic patients admitted to the intensive care unit of an academic hospital. The mitoPO2 will be measured on prespecified measurement moments in the ICU. With each measurement moment, arterial and central venous blood gasses will be taken too.

DETAILED DESCRIPTION:
Evidence is increasing that there is no clear parameter for tissue oxygenation in critically ill septic patients to guide resuscitation. New studies have shown the potential of protoporphyrin IX-triple state lifetime technique to measure mitochondrial oxygenation tension (mitoPO2) in vivo, which possibly is an early indicator of oxygen disbalance in the cell and therefore a physiological trigger for fluid therapy.

Objectives: 1. To describe mitoPO2 measurements in patients with sepsis who are about to receive fluid therapy 2. To describe the effects of fluid therapy and the associated change in mitoPO2 and change in other physiologic measures of tissue oxygenation and oxygen balance 3.To describe the association between mitoPO2 and vital organ (dis)functions and change of SOFA (Sequential organ failure assessment) score after 24hrs 5. To describe the microcirculatory, cellular and mitochondrial function during the first 24 hours of septic patients.

Study population: critically ill patients with sepsis which are admitted to the intensive care unit through the emergency department or hospital ward and in whom fluid therapy (crystalloid, albumin and red cell transfusion) is planned.

Main study endpoints

Primary endpoint: Change in mitoPO2 after fluid therapy. This will be compared to traditional parameters used to measure oxygenation and oxygen balance

Secondary endpoints:

* Association of mitoPO2 trend with separate (ischemic) organ (dis)function. The SOFA score after 24 hours will also be assessed.
* Safety of mitoPO2 measurements in critically ill septic patients.
* Description of the association of sepsis with microcirculatory function, cellular function and mitochondrial function.
* Description of the association between mitoPO2 change and clinical outcomes , like length of stay(both ICU and in-hospital) and mortality (both ICU and in-hospital).

ELIGIBILITY:
Inclusion Criteria:

* Age of patient is at least 18 years
* Patients diagnosed with sepsis in the emergency department or hospital ward
* Patients are admitted to the ICU via the hospital ward or emergency department
* Informed consent is given either by the patient or if the patient is too ill to give informed consent, by his or her legal representative.
* Patients have an arterial catheter in situ, since blood samples will be taken for the study. Most patients admitted to the ICU have an arterial catheter in place since it is part of standard care.

Exclusion Criteria:

* Patients younger than 18 years
* Patients with sepsis discharged after emergency department visit
* Patients admitted to a hospital ward other than the ICU after emergency department visit
* Patients who cannot give informed consent themselves and without a legal representative will be excluded since no informed consent can be obtained
* Patients known with porphyria and/or photodermatosis will be excluded, since the risk of phototoxicity
* Patients with hypersensitivity to the active substance or to the plaster material of ALA (5-aminolevulinic acid)
* Pregnant or breast feeding women since there is no adequate data form the use of ALA in pregnant or breast feeding women
* Insufficient comprehensibility of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the emergency department or hospital ward admitted to the Intensive Care Unit of the Leiden University Medical Center with (the suspicion of) sepsis will be the source population of the study. Leiden Univesity Medical Center is an academic hospital.
  Septic patients are identified as specified in the Dutch protocol of sepsis identification and management in the emergency department. It consists of having clinical suspicion of sepsis in combination with the at least 2 of the following symptoms: ≥ 20 breaths per minute, heart frequency > 90 beats per minute, leukocytes > 12x109 or leukocytes < 4x10^9, and/or temperature > 38 °C or <36 °C
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Change of mitoPO2 during first 24 hours of a septic patient | 24 hours
  The primary endpoint is the change of mitoPO2(mitochondrial oxygenation) before and after fluid therapy in patients with sepsis. This will be compared to traditional parameters used to measure tissue oxygenation and oxygen balance (central venous oxygen saturation, mean arterial pressure and lactate).

SECONDARY OUTCOMES:
SOFA (sequential organ failure assessment) score after 24 hours | 24 hours
  The association of mitoPO2 change in 24 hours with the Sequential Organ Failure Assessment score after 24 hours will be assessed. With the help of this information, more insight can be given in how much information the cutaneous mitoPO2 measurement gives about the organs separately and together.
Organ (dis)function | 24 hours
  To describe the association between mitoPO2 change and separate organ functions.
Validation of mitoPO2 measurement with blood based biomarkers of cellular function | 24 hours
  Cellular function will be assessed with blood-based biomarkers mitochondrial membrane potential (MMP), presence of cellular reactive oxygen species (ROS) molecules and glutathione (GSH) activity. Mitochondrial function will be assessed with mitoPO2 measurements.
Safety (incidence of adverse and serious adverse events) | 24 hours
  The adverse and serious adverse events of the mitoPO2 measurements will be assessed.
Length of ICU stay | 3 months
  Association of mitoPO2 change and length of intensive care unit-stay.
Length of hospital stay | 3 months
  Association of mitoPO2 change and length of hospital stay.
ICU mortality | 3 months
  Association of mitoPO2 change and intensive care unit mortality.
In-hospital mortality | 3 months
  Association of mitoPO2 change and in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna G van der Bom, MD, PhD, Principal Investigator — Leiden University Medical Center; M S Arbous, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No